CLINICAL TRIAL: NCT04860024
Title: The Prospective Role of Epigenetics in Attention-deficit/Hyperactivity Disorderdeficit/Hyperactivity Disorder
Brief Title: Epigenetics in ADHD
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Liang-Jen, Associate Professor and Visiting Staff, Chang Gung Memorial Hospital
Other Study IDs: 104-3522C
Record Dates: First submitted 2021-04-23; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: microRNAs in Attention-deficit/Hyperactivity Disorder
Keywords: attention-deficit/hyperactivity disorder; epigenetics; behavioral science; cognitive function; child and adolescent psychiatry
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We hypothesize that miRNAs' expressions correlate significantly with the phenotypes and neurocognitive endophenotypes of ADHD
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD: Blood sample for miRNA qRT-PCR
  Behavioral and neuropsychological assessments
- Healthy: Blood sample for miRNA qRT-PCR
  Behavioral and neuropsychological assessments

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is among the most common psychiatric disorders in children and adolescents. ADHD's nosology is largely based on clinical phenomenology that includes such symptoms as inattention, hyperactivity and impulsivity. However, a reliable ADHD biomarker has still not been determined either for differential diagnosis or for monitoring treatment effects. MicroRNAs (miRNAs) are small non-coding RNA molecules that function in the process of RNA silencing and the post-transcriptional regulation of gene expression. MiRNAs are found in abundance throughout the nervous system and play a vital role in the transcriptional networks with regards to human brain development. Currently, miRNAs' involvement in the pathogenesis of ADHD continues to be unclear. Therefore, this study aims to investigate the prospective role of miRNAs in ADHD and to determine whether miRNA levels in peripheral blood can serve as a biomarker and a diagnosis panel for ADHD.

In the preliminary study, blood samples were collected from five patients with ADHD and five healthy control subjects. The use of Next Generation Sequencing (NGS) techniques has identified 23 miRNAs as potential biomarkers for ADHD. During this three-year proposal, we intend to recruit 100 drug-naïve patients with ADHD and 100 age- and gender-matched control subjects (Training Set). Blood will be obtained through direct puncture of the vein from each participant to analyze the miRNAs by using quantitative reverse transcription polymerase chain reaction (qRT-PCR). The behavior and neuropsychology of each participant will be assessed. This research will construct a miRNAs diagnosis panel using the Support Vector Machine (SVM) classification model to discriminate ADHD from non-ADHD. The validity of the miRNA diagnosis panel will then be re-examined using an independent validation sample composed of 50 patients with ADHD and 50 control subjects (Testing Set). All of the 150 patients with ADHD will receive treatment in a traditional clinical practice and then will be followed up with for 12 months. At the twelfth month, the same procedures as those performed at the baseline will be replicated to examine the influence of ADHD medications on miRNAs, as well as determine whether miRNAs can serve as a biomarker to portray the condition of ADHD under treatment. MiRNA target gene prediction and functional annotation analysis will also be performed.

This study will develop a potential diagnostic panel for ADHD through the use of combinations of multiple miRNA expressions. We will provide proof of the relationships of miRNAs profiles and ADHD manifestations in clinical samples and further explain the molecular pathogenesis of ADHD. Such information may become an important reference for future research and clinical treatments for patients with ADHD.

DETAILED DESCRIPTION:
Year 1: Recruiting 100 ADHD patients and 100 healthy control subjects (Training Set) to develop a miRNA diagnosis panel for ADHD

1. One hundred eligible ADHD patients that are being treated in the Outpatient Department of Child Psychiatry at Kaohsiung Chang Gung Memorial Hospital in Taiwan will be recruited for this study. One hundred age- and gender-matched control subjects will be found in the same catchment area as that of the patients. After obtaining informed consent from their parents or guardians, research psychiatrists shall interview the participants using the K-SADS-E to confirm the diagnosis. The participants will also undergo WISC-IV assessment to exclude intellectual disabilities.

2. For both the ADHD patients and the healthy control subjects, experienced child psychologists will administer Conners CPT and Conners CATA testing in a room designed to reduce inconsistent testing conditions. Parents or guardians will be required to complete the SNAP-IV parent form and the SAICA; patients' teachers will be required to fill out the SNAP-IV teacher form; and the ADHD-RS and the CGI will be completed and rated, respectively, by a child psychiatrist.

3. Venous blood will be collected from each participant in an EDTA anticoagulant tube. The blood samples will be further processed with the mirVana miRNA isolation kit (Life technology) to extract total RNAs. Based on the preliminary findings, the ΔCt values of the 22 candidate miRNAs will be determined for the 100 ADHD samples and 100 control samples. Then the 10 miRNAs with the smallest p-value will be chosen to develop a miRNAs diagnosis panel for ADHD in the second year.

4. The ADHD patients and healthy control subjects will have 12 months of follow-up. The treatment procedures during that time for patients with ADHD will be determined by the patients' psychiatrists' traditional practice and the agreement of patients and their parents.

1. ADHD patients who decide to receive medical treatment will be prescribed oral short-acting MPH (MPH-IR) two or three times daily, with each dose ranging between 0.3 and 1.0 mg/kg, which shall be determined based on the severity of their clinical symptoms, as well as their age, height, and body weight.
2. The dosage will be adjusted every two weeks to properly improve ADHD symptoms. Changes to long-acting MPH (Ritalin-LA) or extended-release methylphenidate (Concerta) are permitted depending on clinical requirements. The maximum doses of MPH-IR and Ritalin-LA per day are 60 mg and of Concerta is 54 mg, as these are the maximum daily doses approved in Taiwan. The dose will be decreased should any clinically intolerable adverse conditions arise. The final titration dose of MPH with an acceptable response will be maintained through the follow-up period.
3. Concomitant medications are prohibited. Compliance with the drug regimen will be verified at each visit based on reports by the patients' parents and how much of the prescription remains. Patients that start a new medication between the different time-points of the study will be considered dropouts.
4. The ADHD Patients that decide not to receive medical treatment are usually reassessed by a child psychiatrist in the outpatient department once a month and may receive behavioral therapy or re-educative psychotherapy for the duration of the study.
5. The healthy control subjects will be assessed only once, at the baseline. 5. Patients with ADHD will be reassessed at the twelfth month after baseline. The assessment procedures, including miRNAs analysis and ADHD measures, that were administered at baseline will be replicated.

Year 2: Developing a SVM classification model and enrolling an independent validation group with 50 ADHD patients and 50 healthy control subjects (Testing Set)

1. Based on the samples already gathered, the 10 most differentially expressed miRNAs between the ADHD group and control group can be determined. Those 10 values can be used to derive the SVM classification model and create a dependable and strong miRNA diagnosis panel for ADHD. Receiver operating characteristic (ROC) curves will be applied to evaluate the validity of this miRNA diagnosis panel. Both the specificity and sensitivity of this panel are expected to reach 80%.
2. For the independent validation group (Testing Set), 50 eligible patients with ADHD and 50 age- and gender-matched healthy control subjects will be recruited. Research psychiatrists will interview the participants using the K-SADS-E to confirm the diagnosis, and the participants will also undergo WISC-IV assessment to exclude intellectual disabilities.
3. All ADHD patients and healthy control subjects will have experienced child psychologists administer Conners' CPT and Conners' CATA testing. The parents or guardians of the participants are required to complete the SNAP-IV parent form and the SAICA; the patient' teachers are required to complete the SNAP-IV teacher form; and the ADHD-RS and the CGI will be completed and rated, respectively, by a child psychiatrist.
4. Venous blood will be collected from each participant using an EDTA anticoagulant tube. The blood samples will be further processed with the mirVana miRNA isolation kit (Life technology) to extract total RNAs. The levels of the 10 miRNAs elected for the SVM classification model will be determined by qRT-PCR.
5. To verify the results of the Training Set, the miRNAs data of the Testing Set (both the 50 ADHD patients and the 50 healthy control subjects) will be used for blind testing by the miRNA diagnosis panel. The discrimination validity expects both the sensitivity and specificity to reach 80%.
6. The treatment and follow-up procedure for ADHD patients will be the same as in the first year. The 100 ADHD patients recruited in the first year will be followed and reevaluated

Year 3: Completion of the 12-month follow-up of ADHD patients and performing analysis of target genes and enrichment pathways of the miRNAs

1. No new participants will be recruited in the third year. The 12-month follow-up of all 150 patients with ADHD will be completed during this year.
2. The second assessment of patients with ADHD will be carried out to conclude this study (twelfth month after baseline). The same assessment procedures that were administered at baseline will be replicated.

(1) Blood samples will be collected and be processed again to extract miRNAs-. (2) A research psychiatrist will interview the ADHD patients using the K-SADS-E in order to confirm that the patients still meet the diagnostic criteria of ADHD.

(3) Patients with ADHD will undergo neuropsychological testing (WISC-IV, Conners CPT and Conners CATA) and have their behavioral symptoms rated (SNAP-IV, SAICA, ADHD-RS and CGI) by the same rater at baseline. To avoid any bias derived from medication, ADHD patients will be told not to take their medication on the day of the neuropsychological assessment.

3. The trends of the miRNA levels during the 12-month follow-up will be identified. The differential miRNA levels between patients with versus without MPH treatment and between patients who continue versus those who remit from the ADHD diagnosis will be evaluated. Whether miRNAs can function as a biomarker that portrays the ADHD condition after treatment will be determined.

4. The predicted target genes and their enrichment pathways of the differentially expressed miRNAs will be obtained using TargetScan v6.2, miRWalk, and DIANA-microT. The search will focus exclusively on the 3'-UTR regions of the target miRNAs with a p-value of 0.05 defining the probability distribution of random matches set in the software with a minimum miRNA seed length of 7.

ELIGIBILITY:
ADHD

Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition
* The diagnosis of each child had to be made by a child psychiatrist in a structured interview that employed the Kiddie Epidemiologic Version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

Exclusion Criteria:

* History of neuropsychiatric diseases
* Any known major physical illnesses
* Taken any medication to treat ADHD

Health

Inclusion Criteria:

* Age- and gender-matched children without ADHD

Exclusion Criteria:

* History of neuropsychiatric diseases
* Any known major physical illnesses

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Patients with ADHD will be recruited from the out-patient department in Kaohsiung Chang Gung Memorial Hospital, Kaohsiung city, Taiwan
  2. Healthy controls will be recruited from the staff in Kaohsiung Chang Gung Memorial Hospital and from the communities in Kaohsiung city, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
miRNAs | 10 min
  Preliminary results of 23 candidate miRNAs that can function as biomarkers identified by the NGS technique

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, MD, MPH, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Taiwan